CLINICAL TRIAL: NCT05041101
Title: Phase Ib/II Study of Grapiprant (IK-007) and Eribulin Combination Treatment for Metastatic Inflammatory Breast Cancer (mIBC)
Brief Title: Grapiprant and Eribulin for the Treatment of Metastatic Inflammatory Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Termination was requested by study supporter IKENA oncology
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0077; NCI-2021-09158 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0077 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Breast Inflammatory Carcinoma; Recurrent Breast Inflammatory Carcinoma; Stage IV Breast Inflammatory Carcinoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — eribulin; grapiprant; caficrestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (grapiprant, eribulin mesylate) (Experimental): Patients receive grapiprant PO BID on day 1-21 and eribulin mesylate IV over 5 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate; Drug: Grapiprant

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526; Halaven; Halichondrin B Analog
Drug: Grapiprant — Given PO
  Other Names: AAT-007; AT-001; CJ 023,423; CJ-023,423; CJ023,423; RQ-00000007; RQ-07

SUMMARY:
This phase Ib/II trial tests the safety and side effects of grapiprant and eribulin and whether they work to shrink tumors in patients with inflammatory breast cancer that has spread to other places in the body (metastatic). Grapiprant is an anti-inflammatory drug that may prevent tumor growth. Eribulin may block tumor cell growth by stopping tumor cell division. Giving grapiprant and eribulin together may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and efficacy of grapiprant and eribulin combination treatment for the patient with metastatic inflammatory breast cancer (mIBC).

SECONDARY OBJECTIVES:

I. To determine objective response rate (ORR), % of the patients who achieve complete response (CR) or partial response (PR).

II. To determine the time to progression (TTP) of the proposed treatment. III. To determine the duration of response of the proposed treatment. (Phase 2 only) IV. To determine the time to first response of the proposed treatment. (Phase 2 only) V. To determine progression-free survival (PFS) of the proposed treatment. VI. To determine the overall survival (OS) of the proposed treatment. VII. To investigate the predictive biomarker of the proposed treatment.

EXPLORATORY OBJECTIVE:

I. To evaluate the changes in the tumor microenvironment after the proposed treatment.

OUTLINE:

Patients receive grapiprant orally (PO) twice daily (BID) on day 1-21 and eribulin mesylate intravenously (IV) over 5 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age
* Is willing and able to provide written informed consent for the trial
* Has histological confirmation of breast carcinoma with a clinical diagnosis of IBC based on the presence of inflammatory changes in the involved breast, including diffuse erythema and edema (peau d'orange), with or without an underlying palpable mass involving the majority of the skin of the breast. Or the diagnosis confirmed by the MD Anderson IBC specialists. Pathological evidence of dermal lymphatic invasion should be noted but is not required for the diagnosis of IBC
* Any prior treatments will be allowed except eribulin and/or any EP2/4 inhibitor
* Has at least 2 weeks of untreated period from the previous treatment
* Any receptor status for ER/PR and HER2. But for HER2+ type, must has failed trastuzumab, pertuzumab, and T-DM1 treatment.

  * NOTE: HER2 positive status is defined as strongly positive (3+) staining score by immunohistochemistry (IHC), or gene amplification using fluorescence in situ hybridization (FISH), if performed. If IHC is equivocal (2+). HER2 negative status, which is determined by assays using IHC require negative (0 or 1+) staining score. If IHC is equivocal (2+) staining score
* Has a measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 (only applies to phase II part)

  * NOTE: Measurable disease: Measurable lesions are defined as those that can be accurately measured in at least one-dimension (longest diameter to be recorded) as >= 20 mm by chest X-ray, >= 10 mm by computed tomography (CT) scan, >= 10 mm with calipers by clinical exam. Measurable malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be >= 15mm in short axis when assessed by CT scan. Non-measurable disease: All other lesions (or sites of disease), including small lesions, are considered non-measurable. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis, cutis/pulmonitis, inflammatory breast disease, and abdominal masses (not followed by CT or magnetic resonance imaging [MRI]) are considered non-measurable
* Has a distant metastasis site or locoregional recurrence
* Is willing to provide fresh tumor tissue via tumor biopsy before the first dose of the study drug only if participant has a disease can be be safely accessed through a CT-guided/ultrasound (US)-guided or percutaneous biopsy for multiple core biopsies judged by the investigator. If participant doesn't have a disease that can be safely accessed, they are still eligible
* Performance status (PS) of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,200 /mcL
* Platelets >= 100,000 /mcL
* Hemoglobin (Hgb) >= 9 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (up to =< 3 x ULN for patients with liver metastasis)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (up to =< 5 x ULN for patients with liver metastasis)
* Cockcroft-Gault glomerular filtration rate (GFR) (mL/min/1.73 m^2) >= 50
* Left ventricular ejection fraction (LVEF) >= 50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
* Female patients must not be pregnant or breastfeeding and must be practicing a medically acceptable form of locally approved birth control, be sterile or post-menopausal. Male patients should be using a medically acceptable form of birth control during the trial or be sterile

  * Female patient: A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) OR
    * A WOCBP agrees to follow the contraceptive guidance during the treatment period and at least 6 months after the last dose of trial intervention and must refrain from breastfeeding for at least 2 months after the last grapiprant treatment
    * WOCPB must have a negative urine pregnancy test no more than 7 days prior to starting treatment on-study
  * Male patients: A male patient must agree to use contraception during the treatment period and for at least 6 months after the last grapiuprant treatment and refrain from donating sperm during this period
* Patient with human immunodeficiency virus (HIV) including current or prior infection would be included if:

  * With CD4+ T-cell (CD4+) counts >= 350 cells/uL
  * Without a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections

Exclusion Criteria:

* Current chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs), COX-2 inhibitors. We will allow prior use of those agents if patients stop them at least 2 weeks before accrual
* Is currently participating in a study of an investigational anti-cancer agent or receiving concurrent anti-cancer therapy for metastatic disease
* Has a diagnosis of immunodeficiency, or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy
* Uncontrolled hypertension is defined as a systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg, with or without antihypertensive medications
* Has a history of and/or active cardiac diseases

  * History of cardiac diseases including:

    * Active myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular function
    * History of documented chronic heart failure; and documented cardiomyopathy
  * Active cardiac diseases including:

    * Symptomatic angina pectoris within the past 180 days that required the initiation of or increase in anti-anginal medication or other intervention
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with documented compromise in cardiac function
  * Symptomatic pericarditis
* Has preexisting neuropathy > grade 2
* Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative
* Has medical conditions requiring concomitant administration of strong CYP3A4 or P-glycoprotein inhibitors or inducers
* Potentially life-threatening second malignancy requiring systemic treatment within the last 3 years (i.e., patients with a history of prior malignancy are eligible if treatment was completed at least 3 years before entering the Treatment period and the patient has no evidence of disease) or which would impede evaluation of treatment response.
* Hormone ablation therapy is allowed within the last 3 years.
* Patients with history of prior early stage basal/squamous cell skin cancer or non-invasive or in situ cancers that have undergone definitive treatment at any time are eligible.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate if they are stable and have no evidence of new or enlarging brain metastases. They are not using steroids for at least 28 days before trial treatment
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Known active hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Saleem, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 2021~ November 2022. All recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: 8 patients were accrued and assessed for eligibility and 6 patients were assigned to the cohort.
Groups:
- Phase Ib - Dose Level 0: Grapiprant 300 mg BID orally daily, and standard of care eribulin 1.4mg/m2 IV on Day 1 and 8. One cycle is defined as 21 days.
- Phase Ib - Dose Level -1: Grapiprant 200 mg BID orally daily, and standard of care eribulin 1.4mg/m2 IV on Day 1 and 8. One cycle is defined as 21 days.
- Phase II: Recommended Grapiprant Dose (RP2D) from phase Ib and standard of care eribulin 1.4mg/m2 IV on Day 1 and 8. One cycle is defined as 21 days.
Period: Overall Study
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Started | 6 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Diease Progression | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Termination was requested by study supporter IKENA oncology during Phase 1b.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II | Total
Number analyzed (Participants) | 6 | 0 | 0 | 6
Age, Continuous [Median (Full Range); unit: years] | 43 [38 to 56] |  |  | 43 [38 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  |  | 6
  Male | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 1
  Not Hispanic or Latino | 5 |  |  | 5
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 5 |  |  | 5
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 |  |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Determine the Safety of Grapiprant and Eribulin Combination Treatment
Description: Dose-limiting toxicity was defined as probable, possible, and definite events that occurred in the first 21 days (Cycle 1), as prespecified in the protocol.
Time Frame: Up to 21 days from the initial treatment
Population: Termination was requested by study supporter IKENA oncology during Phase 1b.
Measure: Number; unit: participants
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Number analyzed (Participants) | 6 | 0 | 0
participants | 2 |  |

2. Primary Outcome: Determine the Efficacy of Grapiprant and Eribulin Combination Treatment
Description: Clinical Benefit Rate (CBR) was defined as the ratio of patients who achieved a complete response (CR), partial response (PR), or stable disease (SD) (lasting >24 weeks).
Time Frame: Up to 1 year
Population: Termination was requested by study supporter IKENA oncology during Phase 1b.
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Number analyzed (Participants) | 6 | 0 | 0
percentage of participants | 0 |  |

3. Secondary Outcome: Determine Objective Response Rate (ORR)
Description: The percentage of the patients who achieved complete response (CR) or partial response (PR).
Time Frame: Up to 1 year
Population: Termination was requested by study supporter IKENA oncology during Phase 1b.
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Number analyzed (Participants) | 6 | 0 | 0
percentage of participants | 0 |  |

4. Secondary Outcome: Determine the Time to Progression (TTP) of the Proposed Treatment.
Description: Time to progression (TTP), defined as the time from the start of grapiprant treatment to objective tumor progression (PD), was analyzed using the Kaplan-Meier method, and the median with 95% confidence intervals was reported.
Time Frame: Up to 1 year
Population: Termination was requested by study supporter IKENA oncology during Phase 1b.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Number analyzed (Participants) | 6 | 0 | 0
months | 1.54 [1.38 to NA] — Too few subjects remaining at risk beyond the median. Data do not provide enough information to estimate reliable upper CI by using Kaplan-Meier method. |  |

5. Secondary Outcome: Determine the Duration of Response of the Proposed Treatment in Phase II
Description: The time from observing the response to the grapiprant treatment until objective tumor progression (PD)
Time Frame: Up to 2 years
Population: Participants treated at the RP2D in Phase II were intended to be evaluated. However, due to the study's termination during Phase Ib, no participants were analyzed for this objective.
Arm/Group | Phase II
Number analyzed (Participants) | 0

6. Secondary Outcome: Determine the Time to First Response of the Proposed Treatment in Phase II
Description: The time from starting grapiprant treatment until observing the response.
Time Frame: Up to 2 years
Population: as for outcome 5
Arm/Group | Phase II
Number analyzed (Participants) | 0

7. Secondary Outcome: Determine Progression-free Survival (PFS) of the Proposed Treatment
Description: Progression-free survival (PFS) was defined as the time from starting grapiprant treatment until objective tumor progression (PD) or death from any cause and was summarized using the Kaplan-Meier method, including the median with 95% confidence intervals.
Time Frame: Up to 1 year
Population: Termination was requested by study supporter IKENA oncology during Phase 1b.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Number analyzed (Participants) | 6 | 0 | 0
months | 1.54 [1.38 to NA] — Too few subjects remaining at risk beyond the median. Data do not provide enough information to estimate reliable upper CI by using Kaplan-Meier method. |  |

8. Secondary Outcome: Determine the Overall Survival (OS) of the Proposed Treatment
Description: Overall survival (OS) was defined as the time from starting grapiprant treatment until death from any cause and was summarized using the Kaplan-Meier method, including the median with 95% confidence intervals.
Time Frame: Up to 1.5 year
Population: Termination was requested by study supporter IKENA oncology during Phase 1b.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Number analyzed (Participants) | 6 | 0 | 0
months | 10.1 [4.57 to NA] — Too few subjects remaining at risk beyond the median. Data do not provide enough information to estimate reliable upper CI by using Kaplan-Meier method. |  |

9. Secondary Outcome: Investigate the Predictive Biomarker for the Proposed Treatment
Description: Determine the association between treatment response and the change in prostaglandin E2 metabolite (PGEM) levels in urine samples collected pre- and post-treatment.
Time Frame: Baseline and Cycle 2
Population: Patients with treatment response, compared with the non-responder group, were intended to be evaluated for changes in urine PGEM. However, due to the absence of treatment responders in this study, no patients were analyzed for this objective.
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from the initiation of grapiprant treatment through 30 days after the last dose, up to 1 year. All-cause mortality was assessed from the initiation of grapiprant treatment through up to 1.5 years.
Description: Adverse events were assessed according to the CTCAE version 5.0. All study patients who had received any dose of grapiprant were evaluated for safety. Unexpected adverse events, including laboratory adverse events deemed clinically significant by the investigator, were graded and recorded.
Arm/Group | Phase Ib - Dose Level 0 | Phase Ib - Dose Level -1 | Phase II
All-Cause Mortality (participants affected / at risk) | 6/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib - Dose Level 0 (N=6) | Phase Ib - Dose Level -1 (N=0) | Phase II (N=0)
Vomiting (Gastrointestinal disorders) | 1 | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA
Fever (General disorders) | 1 | NA | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | NA | NA
Headache (Nervous system disorders) | 1 | NA | NA
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | NA | NA
Abdominal Pain (Gastrointestinal disorders) | 1 | NA | NA
Skin Infection (Infections and infestations) | 1 | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib - Dose Level 0 (N=6) | Phase Ib - Dose Level -1 (N=0) | Phase II (N=0)
Anemia (Blood and lymphatic system disorders) | 4 | NA | NA
Sinus Tachycardia (Cardiac disorders) | 1 | NA | NA
Abdominal Pain (Gastrointestinal disorders) | 1 | NA | NA
Ascites (Gastrointestinal disorders) | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 2 | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 | NA | NA
Dry Mouth (Gastrointestinal disorders) | 1 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 | NA | NA
Dysphagia (Gastrointestinal disorders) | 1 | NA | NA
Mucositis Oral (Gastrointestinal disorders) | 2 | NA | NA
Nausea (Gastrointestinal disorders) | 2 | NA | NA
Stomach Pain (Gastrointestinal disorders) | 2 | NA | NA
Vomiting (Gastrointestinal disorders) | 2 | NA | NA
Chills (General disorders) | 1 | NA | NA
Edema Limbs (General disorders) | 2 | NA | NA
Fatigue (General disorders) | 1 | NA | NA
Fever (General disorders) | 1 | NA | NA
Pain (General disorders) | 1 | NA | NA
Lung Infection (Infections and infestations) | 1 | NA | NA
Shingles (Infections and infestations) | 1 | NA | NA
Wound Infection (Infections and infestations) | 1 | NA | NA
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | NA | NA
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | NA | NA
Alanine Aminotransferase Increased (Investigations) | 2 | NA | NA
Alkaline Phosphatase Increased (Investigations) | 3 | NA | NA
Aspartate Aminotransferase Increased (Investigations) | 3 | NA | NA
Blood Bicarbonate Decreased (Investigations) | 1 | NA | NA
Blood Bilirubin Increased (Investigations) | 1 | NA | NA
Cardiac Troponin I Increased (Investigations) | 1 | NA | NA
Creatinine Increased (Investigations) | 1 | NA | NA
GGT Increased (Investigations) | 1 | NA | NA
INR Increased (Investigations) | 2 | NA | NA
Lymphocyte Count Decreased (Investigations) | 4 | NA | NA
Lymphocyte Count Increased (Investigations) | 1 | NA | NA
Neutrophil Count Decreased (Investigations) | 2 | NA | NA
Platelet Count Decreased (Investigations) | 1 | NA | NA
Urine Output Decreased (Investigations) | 1 | NA | NA
White Blood Cell Decreased (Investigations) | 5 | NA | NA
Anorexia (Metabolism and nutrition disorders) | 1 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 2 | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 2 | NA | NA
Hyperuricemia (Metabolism and nutrition disorders) | 1 | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 | NA | NA
Hypoglycemia (Metabolism and nutrition disorders) | 1 | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 3 | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 2 | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | NA | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | NA | NA
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | NA | NA
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | NA | NA
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | NA
Aphonia (Nervous system disorders) | 1 | NA | NA
Dizziness (Nervous system disorders) | 1 | NA | NA
Headache (Nervous system disorders) | 1 | NA | NA
Paresthesia (Nervous system disorders) | 1 | NA | NA
Anxiety (Psychiatric disorders) | 2 | NA | NA
Dysuria (Renal and urinary disorders) | 1 | NA | NA
Proteinuria (Renal and urinary disorders) | 1 | NA | NA
Urinary Frequency (Renal and urinary disorders) | 1 | NA | NA
Urine Discoloration (Renal and urinary disorders) | 1 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 3 | NA | NA
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | NA | NA
Hot Flashes (Vascular disorders) | 1 | NA | NA
Hypertension (Vascular disorders) | 4 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT05041101/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT05041101/ICF_000.pdf